CLINICAL TRIAL: NCT07251881
Title: Prospective-randomized Trial to Demonstrate Superiority of SuperCable vs. Conventional Steel Wire for Closure After a Median Sternotomy
Brief Title: SuperCable vs. Conventional Steel Wire for Closure After a Median Sternotomy
Acronym: SURE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-D0040; HumRes67145 (Other: Human Research Switzerland)
Record Dates: First submitted 2025-10-24; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Sternotomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- SuperCable® (Experimental): In the intervention group, sternal closure is performed using the SuperCable® Sternotomy Closure System.
  Interventions: Device: SuperCable®
- Steel wires (Active Comparator): In the control group, sternal closure is performed using conventional USP 7 (United States Pharmacopeia size-designation system) tool steel wires.
  Interventions: Device: Steel Wires

INTERVENTIONS:
Device: SuperCable® — Initially, CABG procedure is performed in standard fashion. In the intervention group, sternal closure is performed using the SuperCable® Sternotomy Closure System.
  Arms: SuperCable®
Device: Steel Wires — Initially, CABG procedure is performed in standard fashion. In the control group, sternal closure is performed using conventional USP 7 (United States Pharmacopeia size-designation system) tool steel wires (Fumedica AG).
  Arms: Steel wires

SUMMARY:
During certain heart surgeries, the sternum is opened and must then be closed securely. The study compares two closure methods - steel wires and SuperCable - in terms of stability, healing, and patient satisfaction. This investigation aims to demonstrate that the iso-elastic properties of the SuperCable Sternal Closure System result in faster sternal bone healing, reduced postoperative pain, shorter hospital stay, and improved physical recovery compared to conventional steel wire sternal closure. Eighty-six patients are participating and are randomly assigned to one of the two groups. After the operation, pain, healing, and possible complications are checked. The patients are examined 3 and 6 months after the operation.

ELIGIBILITY:
Inclusion Criteria:

* Provision of Informed Consent: The subject must have signed and dated the informed consent form prior to any study-related procedures.
* Willingness and Ability to Comply: The subject must express a stated willingness to comply with all study procedures and be available for the duration of the study.
* Age and Sex:

  * Age: The subject must be at least 18 years old.
  * Sex: Both male and female subjects are eligible. In line with the "Sex and Gender in Research Involving Humans" recommendations, data will be stratified and analyzed by sex to identify any potential differences in outcomes.
* Language Competence: The subject must possess sufficient German language skills to accurately complete the postoperative survey
* Travel Capability: The subject must have the ability to travel for all planned study visits, including scheduled CT scans
* Surgical Procedure: The subject must be scheduled for elective coronary artery bypass graft (CABG) procedures, as this is the focus of the investigation
* Adherence to Visit Schedule: The subject must be willing to adhere to all scheduled visits and undergo CT scans as outlined in the study protocol

Exclusion Criteria:

* Pharmacological Restrictions: Current use of corticosteroids or any immunosuppressive medication
* Prior Treatments and Therapies: History of radiation therapy to the thorax
* Reproductive Considerations:

  * Pregnancy, or the intent to become pregnant during the study period
  * Lactation or current breastfeeding
* Allergic Reactions: Known allergic reactions to components of the conventional steel wire or SuperCable, specifically any known metal allergies (e.g., nickel or titanium).

Example: Patients with a documented history of nickel allergy, including previous adverse reactions to products such as sternal cerclages, will be excluded

* Infectious or Febrile Conditions: Any febrile illness occurring immediately before the scheduled surgery
* Concurrent Investigational Treatments: Treatment with another investigational drug or medical device within two months preceding surgery, as well as during the current investigation
* Surgical History: Subjects who have undergone prior sternotomy and osteosynthesis (i.e., re-do patients) will be excluded
* Anatomical Considerations:

  * Known sternal deformities that could compromise the outcome of the investigation
  * Off-midline sternotomy approaches, as these do not align with the surgical technique under investigation
* Patient Residence and Follow-Up Feasibility: Subjects residing in remote regions, including those from interstate or overseas, where follow-up and adherence to the scheduled visits might be compromised
* Other Specific Exclusions: Any additional criteria specific to the disease under investigation or identified by the investigator based on medical judgment (e.g., clinically significant concomitant disease states such as renal failure, hepatic dysfunction, or cardiovascular disease, if these conditions are deemed to interfere with study outcomes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Sternal bone healing | day5, day90, day180 (might be waived depending on outcome on day90)
  Sternal bone healing, assessed via multiplanar CT-scans and a validated quantitative scoring algorithm (Stacy et al., 2014).

SECONDARY OUTCOMES:
Length of Hospital Stay | day90 (Visit 3)
  Length of Hospital Stay is reported
Postoperative pain assessed by using a 10-point visual analog scale (VAS) | day1, day5, day90, day180
  Postoperative pain assessed by using a 10-point visual analog scale (VAS) throughout study. from 0 (no pain) to 10 (most intense pain imaginable)
Total use of opioid-like drugs | day1, day5, day90, day180
  Use of opioid-like drugs is reported using a Pain-Medicine conversion tool, throughout study
Upper Extremity Functional Index Score (UEFI) | day90, day180
  Upper Extremity Functional Index Score (UEFI) is collected. Several items where patients rate their difficulty performing specific activities on a scale from 0 (extreme difficulty) to 4 (no difficulty)
Postoperative Quality of Recovery Scale (PostopQRS) | day90, day180
  Postoperative Quality of Recovery Scale (PostopQRS) is assessed. It is principally comprised of a number of questions that objectively measure patient recovery, which are clustered into five different domains (physiological, emotive, nociceptive, activities of daily living, and cognitive) and one self-assessment domain.
Functional Difficulty Questionnaire (FDQ) | day90, day180
  Functional Difficulty Questionnaire (FDQ) will be conducted
Composite of all complications related to sternal osteosynthesis (i.e., sternal dehiscence, re-operation due to sternal wound healing, wound infections) | day1, day5, day90, day180
  Complications will be collected
Assessment of sternal stability as determined by ultrasound measurement of sternal motion | day5, day90, day180
  Assessment of sternal stability as determined by ultrasound